CLINICAL TRIAL: NCT02789319
Title: DTS Blood Glucose Monitor System Surveillance Program SubStudy 1
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Diabetes Technology Society (Other)
Collaborators: Rainier Clinical Research Center (Other); AMCR Institute (Other); Integrated Medical Development (Industry); Diablo Clinical Research (Unknown); Vanderbilt University Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Diagnostic
Other Study IDs: DTS2016BSP-001-SubSDTS2016-01
Record Dates: First submitted 2016-05-17; First posted 2016-06-03 (Estimated); Last update posted 2018-01-08 (Actual); Status verified 2018-01

CONDITIONS: Diabetes
Keywords: Blood Glucose Monitoring System; BGMS; Diabetes; Patient Use
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (18):
- FreeStyle Lite (Other): Blood Glucose Meter type
  Interventions: Device: Blood Glucose Meter Systems
- Contour Next (Other): Blood Glucose Meter type
  Interventions: Device: Blood Glucose Meter Systems
- OneTouch Ultra2 (Other): Blood Glucose Meter type
  Interventions: Device: Blood Glucose Meter Systems
- ACCU-CHEK AVIVA Plus (Other): Blood Glucose Meter type
  Interventions: Device: Blood Glucose Meter Systems
- Prodigy Auto Code (Other): Blood Glucose Meter type
  Interventions: Device: Blood Glucose Meter Systems
- Walmart ReliOn Prime (Other): Blood Glucose Meter type
  Interventions: Device: Blood Glucose Meter Systems
- Embrace (Other): Blood Glucose Meter type
  Interventions: Device: Blood Glucose Meter Systems
- True Result (Other): Blood Glucose Meter type
  Interventions: Device: Blood Glucose Meter Systems
- True Track (Other): Blood Glucose Meter type
  Interventions: Device: Blood Glucose Meter Systems
- Walmart ReliOn Confirm (Other): Blood Glucose Meter type
  Interventions: Device: Blood Glucose Meter Systems
- Advocate Redi-Code + (Other): Blood Glucose Meter type
  Interventions: Device: Blood Glucose Meter Systems
- CVS Advanced (Other): Blood Glucose Meter type
  Interventions: Device: Blood Glucose Meter Systems
- OneTouch Verio (Other): Blood Glucose Meter type
  Interventions: Device: Blood Glucose Meter Systems
- Contour (Other): Blood Glucose Meter type
  Interventions: Device: Blood Glucose Meter Systems
- Accu-Chek Nano (Other): Blood Glucose Meter type
  Interventions: Device: Blood Glucose Meter Systems
- Walmart ReliOn Ultima (Other): Blood Glucose Meter type
  Interventions: Device: Blood Glucose Meter Systems
- Gmate Smart (Other): Blood Glucose Meter type
  Interventions: Device: Blood Glucose Meter Systems
- SolusV2 (Other): Blood Glucose Meter type
  Interventions: Device: Blood Glucose Meter Systems

INTERVENTIONS:
Device: Blood Glucose Meter Systems

SUMMARY:
The blanket protocol covers the execution of the Diabetes Technology Society (DTS) Blood Glucose Monitor System Surveillance Program that will consist of a series of similar accuracy sub-studies with marketed Blood Glucose Monitor Systems (BGMS) conducted by the Clinical and Laboratory site(s) chosen for this study. The two parts of the study (BGMS testing and comparative glucose analyzer testing) will be conducted in separate facilities (clinical site and laboratory site) so the clinical and laboratory investigators will be blinded from each other's results.

To access the full protocol: http://dst.sagepub.com/content/early/2015/12/10/1932296815614587.full.pdf+html

The clinical site(s) will recruit subjects and test their fingerstick blood directly on the Blood Glucose Monitor Systems. Tubes of fingerstick blood will also be collected from the same subjects, centrifuged and the plasma collected and frozen for shipment to a Clinical Laboratory Improvement Amendments (CLIA)/College of American Pathologists (CAP) certified, accredited clinical chemistry laboratory for measurement on a comparative glucose analyzer. In addition, National Institute of Standards and Technology (NIST) glucose standards (965b) will be assayed on the comparative glucose analyzers to determine any bias from the true glucose values established by the reference mass spectrometry method.

This series of sub-studies will assess the accuracy of various BGMSs by trained professionals, not by the intended end user. Only accuracy of the BGMSs when tests are performed by trained study staff will be assessed. Understanding by the end user of instructions for use (labeling) and human factors analysis are not within the scope of this protocol.

DETAILED DESCRIPTION:
* This is a blanket protocol to cover a series of in vitro diagnostic, Phase 4, sub-studies to determine the performance of 18 various marketed blood glucose meter systems over a 12 month period. All activities performed in these sub-studies will fall within the parameters outlined in this protocol.
* At least 100 and not more than 125 subjects will participate in a sub-study
* All activities will be conducted according to Good Clinical Practice (GCP)
* The protocol, informed consent form, advertisements, and all appropriate documents, will be submitted to an Institutional Review Board (IRB) for approval prior to any study conduct.
* Informed consent will be obtained from each subject for each sub-study. The informed consent form for each sub-study will clearly identify and explain the specific procedures for that sub-study.
* All values obtained by the Blood Glucose Monitor Systems (BGMS) assayed at the clinical site will be compared with glucose values of plasma from the same subjects. Plasma samples will be properly prepared at the clinical site, frozen and shipped on dry ice to a Clinical Laboratory Improvement Amendments (CLIA) /College of American Pathologists (CAP) certified/accredited laboratory for analysis on a glucose comparative instrument
* Glucose Comparative instruments will be tested with appropriate manufacturers controls as well as with National Institute of Standards and Technology (NIST) 965b controls to assure accuracy and quality (analytical imprecision < 2.9% a bias of < 2.2%, and a total error < 6.9%)
* Brief demographic and medical history information will be collected from subjects. In addition, information will be collected regarding medications taken in the previous 48 hours by the subjects such as acetaminophen, ibuprofen, salicylate-containing drugs, ascorbic acid-containing drugs since such compounds could affect the testing results
* Trained study staff will perform both shallow and deep finger punctures on subjects using sterile lancing devices to obtain capillary blood for testing on the BGMSs, as well as for testing on a comparative glucose instrument - subjects will not be asked to do any self-testing
* Subject's capillary blood will be directly applied to the test strip of the BGMSs as per labeling of the device
* In some cases, subject's fingerstick blood will also be collected into a micro-tube and modified (for example, glycolyzed) to obtain blood samples in the hypoglycemic range not BGMSs that are oxygen insensitive since oxygen levels in blood can change during glycolysis.
* Testing of blood may include, but not limited to: -glucose concentration measured on BGMS, hematocrit, comparative glucose assay
* A volume of no greater than 2000 microliters of finger stick capillary blood will be obtained from any subject at a single visit to the site
* No more than ten finger punctures will be performed on any subject. The number and type of finger sticks that a subject may receive in each sub-study will be disclosed in the sub-study informed consent form. All lancets will be sterile; they may either be one time use devices, or lancing device with lancets that are generally used by people with diabetes for self-monitoring of their blood glucose. A new lancing device will be used on each subject.
* Study documents will be retained by the investigative clinical site, the clinical laboratory and Sponsor (Diabetes Technology Society) as required by GCP but no less than 3 years following publication of results.
* Plasma from subjects will be shipped to the accredited clinical laboratory for assay using appropriate shipping methods for biological specimens
* A Contracted Research Organization (CRO) will oversee the studies, monitor the clinical and laboratory sites, conduct Part 11 compliant data management, perform statistical analysis, create reports and post results on clintrials.gov and on the DTS Blood Glucose Monitor System Surveillance Program website that will be created.

To access the full protocol: http://dst.sagepub.com/content/early/2015/12/10/1932296815614587.full.pdf+html

ELIGIBILITY:
Inclusion Criteria:

* Males and females, 18 years of age and older
* People with type 1 or type 2 diabetes, and no diabetes
* At least 66% of subjects will have diabetes
* Approximately 33% of subjects will not have a diagnosis of diabetes (but may have pre-diabetes or previous gestational diabetes)
* Able to speak, read and understand informed consent form in English (unless informed consent forms in other languages become available)

Exclusion Criteria:

* Hemophilia or any other bleeding disorder
* Pregnancy (to eliminate any potential negative effects from the testing procedure on this population, and to reduce liability to the site and sponsor)
* If potential subject has already participated in 4 previous sub-studies in the past 12 months
* A condition, which in the opinion of the investigator or designee, would put the person or study at risk (reason for exclusion will be documented)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1220 (Actual)
Dates: Start 2016-06; Primary Completion 2017-12-31 (Actual); Study Completion 2017-12-31 (Actual)

PRIMARY OUTCOMES:
Analytical accuracy and clinical performance criteria | up to 2 months
  Determine if blood glucose monitoring systems marketed in the US meet pre-determined analytical 199 accuracy and clinical performance criteria. Analytical accuracy/clinical performance criteria were 200 determined by consensus of the DTS BGMS Surveillance Program Steering Committee.

SECONDARY OUTCOMES:
Device issues | up to 2 months
  Obtain data on BGMS device failures or device related problems that may occur during the study

OTHER OUTCOMES:
Results | up to 2 months
  Provide study results to all interested parties through creation of the DTS BGMS Surveillance 205 Website

CONTACTS AND LOCATIONS:
Locations (4):
- United States (4):
  - Diabetes Technology Society, Burlingame, California
  - AMCR Institute, Escondido, California
  - Diablo Clinical Research, Walnut Creek, California
  - Rainier Clinical Research Center, Renton, Washington

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Klonoff DC, Parkes JL, Kovatchev BP, Kerr D, Bevier WC, Brazg RL, Christiansen M, Bailey TS, Nichols JH, Kohn MA. Investigation of the Accuracy of 18 Marketed Blood Glucose Monitors. Diabetes Care. 2018 Aug;41(8):1681-1688. doi: 10.2337/dc17-1960. Epub 2018 Jun 13. PMID 29898901